CLINICAL TRIAL: NCT03624621
Title: RIDEM Integral Remediation for Major Depression. Efficacy Study of a Functional Remediation Program and Cognitive Training
Brief Title: Integral Remediation for Major Depression ("Rehabilitación Integral Para la Depresión Mayor", RIDEM)
Acronym: RIDEM
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospital de Sant Pau (Other)
Collaborators: Instituto de Salud Carlos III (Other Government)
Responsible Party: Principal Investigator, Maria J Portella, Head of the Research Group in Psychiatric Disorders, Hospital de Sant Pau
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: IIBSP-rid-2017-107
Record Dates: First submitted 2018-08-01; First posted 2018-08-10 (Actual); Last update posted 2022-08-30 (Actual); Status verified 2022-08

CONDITIONS: Major Depressive Disorder; Cognitive Symptom
Keywords: Major Depressive Disorder; Cognitive Remediation; Functioning; Full Recovery; Functional Remediation
MeSH Terms: conditions — Depressive Disorder, Major; Neurobehavioral Manifestations | interventions — Cognitive Remediation

STUDY DESIGN:
Intervention Model Description: Randomized single-blind and controlled clinical trial
Who Masked: Outcomes Assessor
Masking Description: Codification of participants, assessor will never know what treatment arm participant was allocated
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Functional Remediation + CCT (Experimental): 12 sessions (1 per week) of group functional remediation program (90 min/session) plus 20 min of tailored computerized cognitive training (CCT)
  Interventions: Behavioral: Functional Remediation; Device: Computerized Cognitive Training (CCT)
- Psychoeducation + Online Games (Placebo Comparator): 12 sessions (1 per week) of psychoeducation for major depression (90 min/session) plus 20 min of playing freely with online games (pre-selected by investigators)
  Interventions: Behavioral: Psychoeducation; Device: Online games
- Treatment as usual (No Intervention): Usual intervention supervised by their psychiatrist

INTERVENTIONS:
Behavioral: Functional Remediation — Functional remediation includes directed group sessions tapping into the main cognitive domains affected in depression (executive functioning, attention and memory) as well as their implication in daily living.
  Other Names: Cognitive Remediation
  Arms: Functional Remediation + CCT
Device: Computerized Cognitive Training (CCT) — 12 add-on sessions (20-minute long) after each group session to train cognitive domains.
  Other Names: CogniFit (registered brand)
  Arms: Functional Remediation + CCT
Behavioral: Psychoeducation — 12 sessions of psychoeducation on depression, providing information about the disease, causes, consequences and other useful data for the management of depression.
  Other Names: Group sessions
  Arms: Psychoeducation + Online Games
Device: Online games — Participants play non-directed online games during 20 minutes after each psychoeducation grup session to make the two active intervention more similar.
  Other Names: friv.com
  Arms: Psychoeducation + Online Games

SUMMARY:
Available pharmacological and psychotherapeutic treatments are not effective for the treatment of cognitive symptoms of major depressive disorder (MDD). More recent studies have described that functional disability and the indirect costs of MDD (e.g., sick leaves at work, decreased productivity, ...) are related to persistent cognitive deficits. Some programs of cognitive rehabilitation and cognitive training (developed for other pathologies) have been tested, but the results are inconsistent.

There is an imperative need to develop a specific comprehensive rehabilitation program for MDD that includes the benefits of traditional functional remediation (FR) and computerized cognitive training (CCT) programs adjusted for each patient's cognitive deficit.

DETAILED DESCRIPTION:
Objectives: To develop the Integral Rehabilitation Program (FR + CCT) and to demonstrate its efficacy in cognitive and functional remission (i.e. global remission) of patients with MDD in clinical remission.

Methodology: The project will consist of two stages:

1. - Development and adaptation of the Integral Rehabilitation program for MD, based on the program developed for bipolar disorder, and including a computerized cognitive training adjusted to the neuropsychological profile of each patient;
2. - A clinical trial, randomized, blind evaluator, with three intervention arms: INTEGRAL REHABILITATION (FR + CCT); PSYCHOEDUCATION + online games; and TREATMENT AS USUAL.

Sample size will be a total of 90 patients with MDD in remission (full or partial).

ELIGIBILITY:
Inclusion Criteria:

* 18 and 60 years (males and females)
* diagnosis of Major Depression (criteria Diagnostic and Statistical Manual 5th edition, DSM-5) in Remission or Partial Remission phase (scores below 14 in the Hamilton Depression Rating Scale-17 items (HDRS-17))
* Cognitive Symptoms (-1.5SD (standar deviation) in objective as subjective tests),
* PDQ > 20
* FAST> 17

Exclusion Criteria:

* Intelligence Quotient (IQ) < 85
* Any medical condition that may affect cognition
* Presence of any comorbid psychiatric condition (including abuse or dependence on substances in the last three months)
* Electroconvulsive therapy (ECT) in the previous year
* Other psychological intervention in the 6 months prior to the study.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 52 (Actual)
Dates: Start 2018-03-15 (Actual); Primary Completion 2020-10-31 (Actual); Study Completion 2020-12-31 (Actual)

PRIMARY OUTCOMES:
Change from baseline Functioning Assessment Short Test (FAST) score at 6 and 15 months | 3 and 12 months after intervention
  Assessment of daily functioning of depressed patients, including economics, cognition, social relationships, leisure and personal care

SECONDARY OUTCOMES:
Change from baseline perceived cognitive deficits (PDQ) | 3 and 12 months after intervention
  Self-appraisal of cognitive functioning

OTHER OUTCOMES:
Change from baseline cognitive functioning | baseline and 12 months after intervention
  Objective neuropsychological battery to assess cognitive domains

CONTACTS AND LOCATIONS:
Overall Officials: Maria J Portella, Dr, Principal Investigator — IBB-Sant Pau
Locations (1):
- Hospital de la Santa Creu i Sant Pau, Barcelona, Catalonia, Spain

IPD SHARING:
Plan to Share IPD: Undecided
Coded database for meta-analysis of cognitive symptoms in MDD (via international consortiums)

REFERENCES:
- [Derived] Vicent-Gil M, Raventos B, Marin-Martinez ED, Gonzalez-Simarro S, Martinez-Aran A, Bonnin CDM, Trujols J, Perez-Blanco J, de Diego-Adelino J, Puigdemont D, Serra-Blasco M, Cardoner N, Portella MJ. Testing the efficacy of INtegral Cognitive REMediation (INCREM) in major depressive disorder: study protocol for a randomized clinical trial. BMC Psychiatry. 2019 May 6;19(1):135. doi: 10.1186/s12888-019-2117-4. PMID 31060604